CLINICAL TRIAL: NCT05402501
Title: Lifestyle Intervention for Patients With Multiple Sclerosis
Acronym: LIMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: National MS Foundation, The Netherlands (Unknown); Voeding Leeft (Unknown)
Responsible Party: Principal Investigator, Ilse Nauta, Coordinating investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2021.0089
Record Dates: First submitted 2022-04-19; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Lifestyle
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple sclerosis (MS): Patients will participate in an online lifestyle program organized by Voeding Leeft, which consists of four main topics: diet, physical activity, relaxation and sleep.
  Interventions: Behavioral: Lifestyle intervention program "Leef! met MS"

INTERVENTIONS:
Behavioral: Lifestyle intervention program "Leef! met MS" — The lifestyle program consists of a three-months intensive program, followed by a 21-months 'inspiration' program with occasional meetings.

SUMMARY:
The LIMS study is an observational study that investigates the effectiveness of an online lifestyle program for patients with multiple sclerosis (MS). The patients will be monitored during 27 months, starting 3 months prior to the start of the lifestyle program.

DETAILED DESCRIPTION:
This study aims to investigate the effect of an online lifestyle program on the impact of multiple sclerosis (MS) on daily functioning. MS patients will participate in the online lifestyle intervention of Voeding Leeft and will complete online questionnaires at 7 time-points: 3 months before the start of the intervention (run-in), before the start of the intervention (baseline), and 3, 6, 12, 18 and 24 months after the start of the intervention. A subsample (n=200) will also take part in measurements through mobile applications. The investigators hypothesize that the lifestyle program will reduce the impact of MS on the patients' daily functioning.

ELIGIBILITY:
Eligibility criteria to participate in the online lifestyle intervention:

Inclusion Criteria:

* MS diagnosis
* Motivated to adapt their lifestyle
* Able to complete online questionnaires by themselves
* Able to do grocery shopping and to (let someone) prepare the meals from the program
* In a subpopulation (n=200): daily use of a smartphone

Exclusion Criteria:

* Not able to participate in an online lifestyle intervention (e.g. not having an email address, laptop/computer, internet)
* An inability to speak or read Dutch
* Vegan diet
* Not willing to eat fish
* BMI <18.5 and >35 kg/m2
* Pregnant or breastfeeding
* Diagnosis of an eating disorder or psychiatric disorder (according to the DSM-V criteria)
* History of bariatric surgery
* Another disorder, such as inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis), cardiovascular disease (e.g. severe heart failure), malignancy, diabetes type 1 and 2
* Having previously participated in a lifestyle intervention of Voeding Leeft or currently participating in another lifestyle program or lifestyle study.
* Currently under treatment at a dietician or lifestyle coach

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis (MS) who signed up for the online lifestyle intervention of Voeding Leeft will be asked to participate in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Impact Scale (MSIS-29) | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures the impact of MS on their daily functioning

SECONDARY OUTCOMES:
12-item Short Form Health Survey (SF-12) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures quality of life
EuroQol 5 Dimensions Questionnaire (EQ-5D) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures quality of life
BMI | Assessed at 7 time-points during 27 months Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  BMI in kg/m^2
Waist circumference | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Waist circumference in centimeters
Bristol stool chart | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Tool used to indicate stool type
Medical Consumption Questionnaire (iMCQ) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures health-care consumption
Hospital Anxiety and Depression Scale (HADS) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures symptoms of depression and anxiety
Checklist Individual Strength-20-r (CIS-20) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures the level of fatigue
Multiple Sclerosis Neuropyschological Screening Questionnaire - patient version (MSNQ-P) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures the level of subjective cognitive complaints
Medical Outcomes Study Sleep Scale (MOS-ss) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures sleep quality
Dutch Norm for Healthy Physical Activity (In Dutch: Nederlandse Norm voor Gezond Bewegen (NNGB)) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures the level of physical activity
Perceived stress scale (PSS) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures the level of perceived stress
iMTA Productivity Cost Questionnaire (iPCQ) | Assessed at 7 time-points during 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Questionnaire that measures work productivity and the frequency of sick leave
Neurokeys keyboard app | Continuous measures during a period of 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Only in a subsample (n=200); Real-world keystroke dynamics collected by smartphone technology.
MS sherpa app - Smartphone-adapted Symbol Digit Modalities Test (sSDMT) | Weekly tests during a period of 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Only in a subsample (n=200); Patients will use the MS sherpa app to perform a smartphone-adapted Symbol Digit Modalities Test (sSDMT) on their mobile phone.
MS sherpa app - Smartphone-adapted two-minute walking test | Weekly tests during a period of 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Only in a subsample (n=200); Patients will use the MS sherpa app to perform a two-minute walking test outside.
MS sherpa app - questionnaire | Weekly questionnaire during a period of 27 months | Change over time between baseline and follow-up time-points will be compared to change over time between the run-in period and baseline.
  Only in a subsample (n=200); Patients will use the MS sherpa app to answer seven questions on a likert-scale (e.g. about pain, stress, energy, memory) within the mobile application.

CONTACTS AND LOCATIONS:
Overall Officials: Brigit de Jong, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided